CLINICAL TRIAL: NCT06804525
Title: Use of Life History Calendars to Enhance Measurement of Lifetime Experience With Mental Disorders in Hong Kong.
Brief Title: LHC-CIDI-5 in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Michael Y. Ni, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW 24-771; 2024-0089-004 (Other Grant/Funding Number: Hong Kong Jockey Club Charities Trust)
Record Dates: First submitted 2025-01-24; First posted 2025-02-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Episode (MDE); Major Depressive Disorder (MDD); Persistent Depressive Disorder (PDD); Suicidal Ideation; Suicidal Plan; Suicidal Attempt; Suicidal Gesture; Nonsuicidal Self-Injury; Manic Episode; Hypomanic; Bipolar I Disorder; Bipolar Sub Disorder; Bipolar II Disorder; Generalized Anxiety Disorder (GAD); Intermittent Explosive Disorder (IED); Panic Attack; Panic Disorder; Obsessive-Compulsive Disorder (OCD); Posttraumatic Stress Disorder (PTSD); PCL-SC PTSD; PCL-5 PTSD; Alcohol Use Disorder (AUD); Substance Use Disorder (SUD)
Keywords: Life History Calendar; CIDI; Recall bias; Retrospective reporting; Lifetime prevalence; Mental disorders
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation; Self-Injurious Behavior; Mania; Bipolar Disorder; Generalized Anxiety Disorder; Disruptive, Impulse Control, and Conduct Disorders; Panic Disorder; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Alcoholism; Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CIDI-5: For the CIDI-5 group, respondents will directly partake in the CIDI-5 interview without responding to any inquiries regarding their life history.
  Interventions: Diagnostic Test: CIDI-5
- LHC-CIDI-5: For the LHC-CIDI-5 group, respondents, before initiating the CIDI-5, will begin with LHC, completing a calendar by answering questions about important personal experiences since birth until the interview year.
  Interventions: Diagnostic Test: LHC-CIDI-5

INTERVENTIONS:
Diagnostic Test: CIDI-5 — The World Health Organization Composite International Diagnostic Interview-5th (CIDI-5) is a standardized diagnostic tool used to assess the prevalence of mental and substance use disorders over varying time frames (30 days, 12 months, and lifetime) based on the diagnostic criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) and International Classification of Diseases 10th edition (ICD-10) . Trained interviewers will administrate selected modules from the Hong Kong version of the CIDI-5 in a computer-assisted personal interview to measure the outcomes.
  Groups: CIDI-5
Diagnostic Test: LHC-CIDI-5 — The interviewer will start by asking the respondent's age and significant personal experiences, which is expected to take 15 minutes. Remembering and recording the experiences provide cognitive engagement and information which can further serve as memory cues for respondents in the following screening of CIDI-5. Subsequently, the respondents will proceed to the screening section for CIDI-5 and will refer to the completed calendar from the LHC section when they are asked to report lifetime experience or age-of-onset for mental disorders. Trained interviewers will conduct all interviews in a computer-assisted personal interview. To validate the diagnoses in the LHC-CIDI-5 group, clinical re-interviews for MDD, GAD, and PTSD will be conducted by a trained mental health professional with previous experience using DSM-5.
  Groups: LHC-CIDI-5

SUMMARY:
The World Health Organization Composite International Diagnostic Interview-5th (CIDI-5) is a standardized diagnostic tool used to assess the prevalence of mental and substance use disorders over varying time frames (30 days, 12 months, and lifetime) based on the diagnostic criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) and International Classification of Diseases 10th edition (ICD-10). However, retrospective measurements like the CIDI-5 are susceptible to recall bias, especially for the lifetime experience, which can hinder the reporting accuracy with mental disorders.

To mitigate this issue, the life history calendar (LHC) was introduced as an aid to assist respondents in recalling the timing of life events, enhancing the ability of the CIDI-5 to measure the lifetime prevalence of mental disorders. The LHC is a grid structure with columns representing time units and rows representing life domains under study.

In a study conducted in Nepal, combining the CIDI-5 with the LHC resulted in a significant increase in the detection of mental disorders compared to using the CIDI-5 alone. This approach did not lead to an increase in false positives after clinical validation.

This experiment aims to adapt a Hong Kong version of the LHC based on the Nepalese model and evaluate the effectiveness of the LHC-assisted CIDI-5 (LHC-CIDI-5) compared to the CIDI-5 alone in assessing mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* All household members aged 25 years old and over are randomly sampled from the Census and Statistics Department List of Quarters
* Live in the address sampled from the Census and Statistics Department List of Quarters
* Reside in Hong Kong for at least six months in the past year
* Able to read and communicate in Chinese or English
* Without linguistic or cognitive difficulties

Exclusion Criteria:

* Domestic workers

Min Age: 25 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a sub-study of the District Health Profile (DHP), which is a district-level representative descriptive cross-sectional study. In DHP, 1% of households in selected Hong Kong districts will be randomly selected from the Census and Statistics Department's list of quarters, with stratification based on districts and housing types; all persons aged 18 and above in the recruited households will be included and surveyed. For participants who consent to join the DHP study, a sub-sample of 2,500 participants aged 25 or above will be randomly selected and assigned to two groups through a random process. All 2,500 individuals will complete the survey for the DHP study, including the CIDI-5 section. When administering the CIDI-5, one group of 1,250 individuals will be interviewed using only the CIDI-5, while the other group of 1,250 individuals will be interviewed with LHC first, followed by the CIDI-5.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Depression | Immediately following intervention or recruitment
  The main outcomes in this module are the lifetime prevalence of Major Depressive Episode (MDE) and Major Depressive Disorder (MDD)
Persistent Depression | Immediately following intervention or recruitment
  The main outcome in this module is the lifetime prevalence of Persistent Depressive Disorder (PDD)
Self Harm | Immediately following intervention or recruitment
  The main outcomes in this module are the lifetime prevalence of Suicidal Ideation, Suicidal Plan, Suicidal Attempt, Suicidal Gesture, and Nonsuicidal Self-Injury.
High Mood | Immediately following intervention or recruitment
  The main outcomes in this module are the lifetime prevalence of Manic Episode, Hypomanic, Bipolar I Disorder, Bipolar Sub Disorder, and Bipolar II Disorder
Worry and Anxiety | Immediately following intervention or recruitment
  The main outcome in this module is the lifetime prevalence of Generalized Anxiety Disorder (GAD)
Anger Attacks | Immediately following intervention or recruitment
  The main outcome in this module is the lifetime prevalence of Intermittent Explosive Disorder (IED)
Panic Attacks | Immediately following intervention or recruitment
  The main outcomes in this module are the lifetime prevalence of Panic Attack and Panic Disorder.
Obsessions and Compulsions | Immediately following intervention or recruitment
  The main outcome in this module is the lifetime prevalence of Obsessive-Compulsive Disorder (OCD)
Stressful Experiences | Immediately following intervention or recruitment
  The main outcomes in this module are the lifetime prevalence of Posttraumatic Stress Disorder (PTSD), PCL-SC PTSD, and PCL-5 PTSD.
Tobacco, Alcohol, and Drugs | Immediately following intervention or recruitment
  The main outcomes in this module are the lifetime prevalence of Alcohol Use Disorder (AUD) and Substance Use Disorder (SUD)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y. Ni, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, SAR, Hong Kong

REFERENCES:
- [Background] Amro I, Ali A, Hassan MHMO, Al Shawwaf M, Alhassan A, Al Bahari D, El Fakki H, Hijawi Z, Aly S, Amin A, Mohammed R, Nofal M, Abdelkader M, Salman S, Currie J, Alabdulla M, Sampson NA, First M, Kessler RC, Woodruff PW, Khaled SM. Design and field procedures for the clinical reappraisal of the Composite International Diagnostic Interview version 3.3 in Qatar's national mental health study. Int J Methods Psychiatr Res. 2023 Sep;32(3):e1958. doi: 10.1002/mpr.1958. Epub 2023 Jan 18. PMID 36654500
- [Background] Axinn WG, Chardoul S, Gatny H, Ghimire DJ, Smoller JW, Zhang Y, Scott KM. Using life history calendars to improve measurement of lifetime experience with mental disorders. Psychol Med. 2020 Feb;50(3):515-522. doi: 10.1017/S0033291719000394. Epub 2019 Mar 11. PMID 30854987